CLINICAL TRIAL: NCT02692690
Title: Electromagnetic Interference by Transcutaneous Neuromuscular Electrical Stimulation in Patients With Optimizer(R) - a Pilot Safety Study
Brief Title: TENS in Optimizer(R) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Wolzt, Prof. MD, Prof Dr Michael Wolzt, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1067_2015
Record Dates: First submitted 2016-01-28; First posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- before-after (Experimental): TENS stimulation neck and thigh
  Interventions: Device: Stimulette r4x

INTERVENTIONS:
Device: Stimulette r4x

SUMMARY:
Systemic skeletal muscle atrophy (cachexia) is a typical side effect of chronic heart failure.

Patients with cachexia can benefit from transcutaneous electrical neuromuscular stimulation (TENS). It is applied to strengthen the musculature and improve exercise tolerance and quality of life.

It is unclear if application of TENS can cause electromagnetic interference (EMI) in patients with Optimizer® pacemaker systems for improvement of heart failure.

This pilot safety study enrolled 6 patients with chronic heart failure and reduced left ventricular ejection fraction. All patients had an Optimizer® pacemaker system implanted for a minimum of 6 months, no patients had any ventricular arrhythmic episode 3 months prior to the study, and all were in clinically stable condition and willing to participate in this study.

Neuromuscular stimulation was administered via TENS in 4 different modes (HF, LF, Burst, MF) on the right and left musculus trapezius and on both musculi quadriceps femoris. All patients were tested for EMI without or with cardiac contractility modulation (CCM) delivery of the Optimizer®-system respectively.

ELIGIBILITY:
Inclusion Criteria:

* >18 years, with implantation of the Optimizer ® >6 months ago, clinically stable condition and without any ventricular arrhythmic episode in the last 3 months.

Exclusion Criteria:

* Local swelling or edema at the site of stimulation, intolerance to electrical stimulation, or presence of other metallic implants at the site of stimulation

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The patients with CCM-system are assessed for EMI during TENS-application | 6 months
  Electromagnetic interference can cause artificial sensing in pacemaker or ICD system. These artefacts may have the effect of suppressing the pacemaker pulses sensing of tachycardia in ICD.
  The patients will be exposed to electrical stimulations, which will be of different forces on the neck and the upper thigh with r4x. These impulses and the effects will be noted down. It will be investigated if there is an interference with the optimizer ® depending on the different sites of the electrical stimulations and the different impulse forces.
  Many patients with an Optimizer ® have simultaneously a pacemaker - or ICD implant. A special extra monitor will note if there are probable interferences with these pacemaker- or ICD implants.

IPD SHARING:
Plan to Share IPD: No